CLINICAL TRIAL: NCT03325309
Title: Barriers and Facilitators to a Home-based Cycling Program Tailored to Patients' Preferences in Lumbar Spinal Stenosis Using Connected Ergometric Bicycles: a 3-month Open Pilot Study
Brief Title: Barriers and Facilitators to Cycling for Lumbar Spinal Stenosis
Acronym: FLEXCAL Pilot
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Université Paris Descartes (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI16029H
Record Dates: First submitted 2017-10-12; First posted 2017-10-30 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2017-10

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar spinal stenosis; Cycling; Lumbar-flexion-based training
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home-based cycling: A single outpatient supervised session followed by a 3-month home-based cycling program tailored to patients' preferences
  Interventions: Other: Home-based cycling

INTERVENTIONS:
Other: Home-based cycling — A single outpatient supervised session followed by a 3-month home-based cycling program tailored to patients' preferences

SUMMARY:
The purpose of this study is to determine whether a home-based cycling program for patients with lumbar spinal stenosis is a feasible and acceptable

DETAILED DESCRIPTION:
Lumbar spinal stenosis is a prevalent and disabling condition in elderly individuals. Lumbar spinal stenosis results in lumbar and/or radicular leg pain when standing and walking, while symptoms regress in lumbar flexion positions and at rest. The inability to stand or walk impairs functioning and health-related quality of life of elders, and has an important healthcare cost. The 2 main treatment options for lumbar spinal stenosis are conservative or surgical. Laminectomy may be more effective on pain and function than conservative therapy. However, the benefit-risk balance of surgery should be considered in this population with numerous co-morbidities, and evidence is inconsistent. Therefore, conservative therapy is usually the first line option to avoid or delay surgery. Data regarding exercise therapy are scarce. Lumbar-flexion-based exercises are usually recommended. A pilot study suggested that lumbar-flexion-based endurance training, namely cycling, could be an effective and safe method to improve pain, function and health-related quality of life in elderly patients with chronic low back pain but barriers to adhering to the program were detected. Investigators aim to assess barriers and facilitators to a 3-month home-based cycling program in lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilment of International Society for the Study of Lumbar Spine clinical diagnosis criteria for lumbar spinal stenosis with the presence of at least 6 out of the 7 following criteria: "pain in the buttocks or legs while walking"; "flex forward to relieve symptoms"; "feel relief when using a shopping cart or bicycle"; "motor or sensory disturbance while walking"; "normal and symmetric foot pulses"; "lower extremity weakness"; and "low back pain"
* Lumbar spinal stenosis qualitatively detected on MRI or CT-scan

Exclusion Criteria:

* Inability to speak or read French
* Impossibility or refusal to have an ergometric bicycle at home
* Ongoing lumbar-flexion-based endurance training
* History of spinal surgery
* Cognitive impairment
* Neurological or vascular disorder involving the lower limbs
* Contraindication to cycling

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 50 year-old with symptoms related to degenerative lumbar spinal stenosis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Barriers to home-based cycling | 3 months
  Assessed by a qualitative approach using semi-structured interviews
Facilitators to home-based cycling | 3 months
  Assessed by a qualitative approach using semi-structured interviews

SECONDARY OUTCOMES:
Barriers to home-based cycling | Baseline
  Assessed by a qualitative approach using semi-structured interviews
Facilitators to home-based cycling | Baseline
  Assessed by a qualitative approach using semi-structured interviews
Number of training sessions to assess adherence to home-based cycling | 3 months
  assessed by automatic monitoring on a USB stick connected to the bicycle
Covered distance to assess adherence to home-based cycling | 3 months
  assessed by automatic monitoring on a USB stick connected to the bicycle
Duration of training sessions to assess adherence to home-based cycling | 3 months
  Number of training sessions, distance, duration and power assessed by automatic monitoring on a USB stick connected to the bicycle
Developed power to assess adherence to home-based cycling | 3 months
  assessed by automatic monitoring on a USB stick connected to the bicycle
Burden of a home-based cycling | 3 months
  Assessed by the Exercise Therapy Burden Questionnaire (0=no burden, and 100=maximal burden)
Mean change from baseline in mean lumbar pain in the past 48 hrs | 3 months
  Assessed by an 11-point numeric rating scale (0=no pan, and 100=maximal pain)
Mean change from baseline in mean radicular pain in the past 48 hrs | 3 months
  Assessed by an 11-point numeric rating scale (0=no pain, and 100=maximal pain)
Mean change from baseline in mean disability in the past 48 hrs | 3 months
  Assessed by an 11-point numeric rating scale (0=no disability, and 100=maximal disability)
Mean change from baseline in mean spine-specific activity limitation | 3 months
  Assessed by the Oswestry Disability Index (0=no limitation, and 100=maximal limitation)
Mean change from baseline in mean maximum walking distance | 3 months
  Assessed by an adapted version of the self-paced walking test

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Nguyen, MD, PhD, Principal Investigator — A_HP
Locations (1):
- Hôpital Cochin -Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pauwels C, Roren A, Gautier A, Linieres J, Rannou F, Poiraudeau S, Nguyen C. Home-based cycling program tailored to older people with lumbar spinal stenosis: Barriers and facilitators. Ann Phys Rehabil Med. 2018 May;61(3):144-150. doi: 10.1016/j.rehab.2018.02.005. Epub 2018 Feb 27. PMID 29499383